CLINICAL TRIAL: NCT00254514
Title: A Multi-centre, Randomised, Double-blind, Placebocontrolled, Parallel-group Trial Investigating the Efficacy and Safety of Norditropin® SimpleXx® in Tibia Fractures
Brief Title: Controlled Study to Evaluate the Efficacy and Safety of the Treatment With Growth Hormone in Tibia Fractures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1606-1365
Record Dates: First submitted 2005-11-15; First posted 2005-11-16 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Bone Fracture; Tibia Fractures
MeSH Terms: conditions — Fractures, Bone | interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: somatropin

SUMMARY:
This trial is conducted in Africa, Europe and Middle East. This trial investigates the efficacy and safety of three dose levels of Norditropin® (growth hormone) as compared to placebo in the treatment of tibia fractures. The trial will be conducted in two parts: in the first part, the patients will be evaluated with regard to efficacy (fracture healing) and safety at short time intervals until week 24 post-surgery. In the second part, long-term safety and fracture healing up to 12 months post-surgery will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Primary surgical treatment of tibia fracture using intramedullary nailing
* Closed fractures: Tscherne Type C1, C2 and C3
* Open fractures: Gustilo Grade I, II and IIIa

Exclusion Criteria:

* Open growth plate on X-rays
* Known chronic endocrine or metabolic disease including diabetes and severe obesity defined as body mass index (BMI)1 > 32.0
* Severe head injury defined as patients who are stuporous or comatose with pupillary enlargement or asymmetry
* Critically ill patients defined as patients in need of mechanical ventilation (except during surgical procedures) or circulatory support (defined as use of inotropic drugs)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2001-08; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Time from surgery until fracture has healed | During a 12 month period

SECONDARY OUTCOMES:
Investigator's assessment: fracture healed
Number of fractures healed

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (35):
- Finland (2):
  - Novo Nordisk Investigational Site, Kuopio
  - Novo Nordisk Investigational Site, Oulu
- Novo Nordisk Investigational Site, Strasbourg, France
- Germany (11):
  - Novo Nordisk Investigational Site, Augsburg
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Braunschweig
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Homburg
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Mainz
  - Novo Nordisk Investigational Site, München
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Offenbach
  - Novo Nordisk Investigational Site, Würzburg
- Hungary (4):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Győr
  - Novo Nordisk Investigational Site, Miskolc
  - Novo Nordisk Investigational Site, Veszprém
- Israel (5):
  - Novo Nordisk Investigational Site, Beersheba
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Kfar Save
  - Novo Nordisk Investigational Site, Tel Aviv
- Norway (2):
  - Novo Nordisk Investigational Site, Lillestrøm
  - Novo Nordisk Investigational Site, Oslo
- Poland (5):
  - Novo Nordisk Investigational Site, Gorzów
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Piekary Śląskie
  - Novo Nordisk Investigational Site, Sosnowiec
  - Novo Nordisk Investigational Site, Szczecin-Zdunowo
- South Africa (3):
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
  - Novo Nordisk Investigational Site, Worcester
- Spain (2):
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Valencia

REFERENCES:
- [Result] Raschke M, Rasmussen MH, Govender S, Segal D, Suntum M, Christiansen JS. Effects of growth hormone in patients with tibial fracture: a randomised, double-blind, placebo-controlled clinical trial. Eur J Endocrinol. 2007 Mar;156(3):341-51. doi: 10.1530/EJE-06-0598. PMID 17322494
- [Derived] Krusenstjerna-Hafstrom T, Rasmussen MH, Raschke M, Govender S, Madsen J, Christiansen JS. Biochemical markers of bone turnover in tibia fracture patients randomly assigned to growth hormone (GH) or placebo injections: Implications for detection of GH abuse. Growth Horm IGF Res. 2011 Dec;21(6):331-5. doi: 10.1016/j.ghir.2011.08.003. Epub 2011 Oct 1. PMID 21963127
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com